CLINICAL TRIAL: NCT02564432
Title: Microbiome and Innate Immunity With Percutaneous Osseointegrated Prostheses
Brief Title: Microbiome and Metagenome in Percutaneous Osseointegrated Prostheses (MMPOP)
Acronym: MMPOP
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: A1544-I
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Transfemoral Amputation
Keywords: amputee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stomal and skin swab samples for bacterial 16S ribosomal RNA and fungal 18S ribosomal RNA. Blood samples to detect messenger ribonucleic acid (mRNA) of genes regulating production of immune proteins. Serous drainage from the stoma to determine wound healing cytokine expression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- POP 10 patient cohort: This is an observational study

SUMMARY:
The purpose of this study is to investigate the clinical implementation of a new percutaneous prosthetic attachment system by determining the resident microbial ecology of the implant exit site and to simultaneously study the systemic and local stomal immune responses. This study will follow 10 patients implanted with percutaneous osseointegrated prosthetics (POPs) for a period of one year. Two state-of-the-art, pre- and post-surgery bacterial monitoring technologies will be used; these procedures are intended to facilitate the early prediction, detection, and treatment of infection, as well as to provide follow-up data that can potentially be used to advantageously manipulate the stomal microbial environment in future clinical trials.

Commensal skin bacteria colonize all stomas. Colonization does not necessarily result in infection. Over time, the presence of this skin penetrating foreign object (implant) will cause measurable changes in the bacterial population (microbiota) at and around the POP exit site. It is anticipated that the evolving microbiota, in concert with measurable changes in the local and systemic cytokine responses, will reveal patterns associated with mutualistic-commensal bacteria and/or pathogenic bacteria related to the stages of chronic wound healing. These patterns could be used to determine the presence of a stable uninfected stoma or the progression of a stomal infection. Hopefully, this information will allow timely intervention to prevent infection, i.e. by detecting early stages of infection or discerning common patterns of stable mutualistic-commensal bacterial strains, effective intervention protocols (antibiotics, probiotics or manipulation of the stomal and skin microbiota) may be developed to avoid patient morbidity and assure implant survival.

DETAILED DESCRIPTION:
Percutaneous osseointegrated prosthetic (POP) attachment (i.e., the direct skeletal attachment of artificial limbs) is a rapidly evolving technology. This follows over a decade of successful European trials that largely involved transfemoral amputees. This information together with the translational animal studies have made it possible to commence an Early Feasibility Device Exemption (IDE) Pilot Program under the direction of the Federal Drug Administration (FDA). Ten transfemoral amputees, selected from the Veteran and active military populations will receive a novel POP device. The objective of this study is to follow 10 patients implanted with a POP for a period of one year.

All stomas are colonized by local skin bacteria; colonization does not necessarily result in infection. Over time, the presence of this skin penetrating foreign object (implant) will cause measurable changes in the bacterial population (microbiota) at and around the POP exit site.

It is anticipated that the evolving microbiota, in concert with measurable changes in the local and systemic cytokine responses, will reveal patterns associated with mutualistic-commensal bacteria and/or pathogenic bacteria related to the stages of chronic wound healing. These patterns could be used to determine the presence of a stable uninfected stoma or the progression of a stomal infection. Hopefully, this information will allow timely intervention to prevent infection, i.e. by detecting early stages of infection or discerning common patterns of stable mutualistic-commensal bacterial strains, effective intervention protocols (antibiotics, probiotics or manipulation of the stomal and skin microbiota) may be developed to avoid patient morbidity and assure implant survival.

The study aims will test the following:

Aim 1: Determine and characterize the microbiota in the region surrounding the skin/implant interface. Sampling will take place over all stages of wound healing and stomal maturation and will begin with Stage 1 and Stage 2 surgeries, as well as at defined time points, and collection sites (i.e., the stoma, ipsilateral and contralateral thigh skin) for up to one year post surgery. This will be carried-out by using a specific swabbing technique to collect bacterial and fungal deoxyribonucleic acid (DNA) and to amplify and sequence bacterial 16 Svedberg units ribosomal ribonucleic acid (16S rRNA) and fungal 18 Svedberg units ribosomal ribonucleic acid (18S rRNA) genes.

AIM 2: Compare the expression patterns of the local and systemic inflammatory biomarkers over time and determine if there is a correlation with the microbiota pattern to diagnose the state of wound healing at the skin/implant interface and the systemic response to a potentially life-long chronic wound. The measurements of the pro-inflammatory cytokines, found in the stomal exudate (local biomarkers) and blood serum (systemic biomarkers), along with evolving microbiota profiles (Aim #1) will help to better characterize the homeostatic state of the stoma and subsequent optimum wound care therapies.

The ability to predict infection and to avoid it without the use of antibiotics would be of great value to future clinical trials. Assuming the success of this feasibility pilot trial, it is anticipated that the trial will be expanded to include 200 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Is a US military Veteran with transfemoral limb loss, that occurred at least 6 months prior to consent, and that the amputation is not a result of dysvascular disease.
2. Is at least 18 years of age or older.
3. Has previously used or is currently using a "socket suspension technology" prosthesis
4. Has, in the opinion of the investigator, normal cognitive function and no physical limitations, addictive diseases, or underlying medical conditions including tobacco use (continued testing for tobacco use will be performed at screening) that may prevent the subject from being an appropriate study candidate.
5. Is willing, able, and committed to participation in baseline and follow-up evaluations for the entire duration of the study.
6. Can provide written informed consent to participate.

Exclusion Criteria:

1. Is currently on active or reserve military duty
2. Has experienced systemic bacterial infection or localized infection at the stump site within the previous 6 months
3. Has had more than 1 limb amputated
4. Has a body mass index (BMI) 30
5. Has insulin dependent diabetes mellitus (IDDM) or has adult onset DM with a glycated hemoglobin (HbA1c) > 53 mmol/mol (7.0%) at screening
6. Has residual femur bone length of less than 25% of the length of the contralateral femur.
7. Has clinically diagnosed vascular compromise proximal to the surgical site
8. Is pregnant at the time of surgery or plans to become pregnant within the first year of follow-up
9. Has evidence of recent tobacco use (urine cotinine test > 300 ng/mL [1703 nmol/L]) and is not committed to a smoking-cessation program
10. Has renal insufficiency (defined as serum creatinine of 1.8 mg/dL) or is currently receiving renal dialysis
11. Is currently involved in or plans to be involved in high levels of physical activity (competitive sports, heavy physical labor, etc) during the first 12 months of the rehabilitation stage
12. Has muscular, neurologic or vascular deficiencies that may compromise the bone or soft tissue healing of the affected extremity
13. Has anemia characterized by a hemoglobin of 11 g/dL at the time of surgery
14. Is currently on oral anticoagulation (excluding low-dose aspirin for cardiac prophylaxis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 transfemoral amputees selected from Veteran and active military populations
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P Beck, MD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients, who were recruited to participate in the early feasibility study of the percutaneous osseointegrated prosthesis (NCT02720159), were also recruited to participate in this study. Patients were transfemoral amputees selected from the VA patient registry
Groups:
- Stomal and Skin Microbiota: Unilateral transfemoral amputees, who were fitted with a single percutaneous osseointegrated prosthetic device, were included in this study. The microbiota of the stoma (the skin exit site through which the percutaneous post protrudes) was sampled at defined time points for 16S (Svedberg unit) rRNA (ribosomal ribonucleic acid) and followed for 12 months, after the Stage 2-surgery. Microbiota from each patient's healthy ipsilateral thigh skin were used as controls. Thus, each patient had an internal control at each sampling point.
Period: Overall Study
Arm/Group | Stomal and Skin Microbiota
Started | 10
Completed | 8 (1 patient suffered periprosthetic fracture at 8 months; 1 failed to osseointegrate)
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- POP 10 Patient Cohort: Patient who are fitted with POP devices
Arm/Group | POP 10 Patient Cohort
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Fitted with a percutaneous osseointegrated prosthesis [Number; unit: Number of patients] | 10

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Community Types as Determined by Percentage RNA Sequence Reads
Description: To compare, within each participant, the Bacterial Community Type dynamics over time, we used Loess regression to visualize local (temporal) trends in the data. Specifically, it takes the scatter-plot of values (relative abundances, diversity indices) and uses smoothing to identify local trends in the data. As percentage RNA sequence reads were the measure of central tendency, measure of dispersion of the data was not possible to calculate.
Time Frame: On Day 3 after first surgery and day 3 prior to and days, 3, 14 and week 6 and months 3, 6, 9 and 12 after second surgery.
Population: Microbiota from implant stoma and ipsilateral thigh skin.
Measure: Number; unit: Percentage RNA sequence reads
Groups:
- Stoma Microbiota: Patients implanted with POP devices
- Healthy Thigh Skin Microbiota: Patient's thigh skin with and without POP implants (which proved to be the same and the ipsilateral thigh skin was used for final analysis)
Arm/Group | Stoma Microbiota | Healthy Thigh Skin Microbiota
Number analyzed (Participants) | 10 | 10
Percentage RNA sequence reads
  Staphylococcus | 3.4 | 4.6
  Streptococcus | 4.7 | 8.7
  Corynebacterium | 2.2 | 24.0
Statistical Analysis 1: Comparison: Stoma Microbiota vs Healthy Thigh Skin Microbiota; Sample similarity was calculated using the statistical comparisons of community composition; Test type: Equivalence — This is not a randomized clinical trial but is an observational study, each patient's thigh skin site served as the control; p < 0.05, Unweighted UniFrac (qualitative) — The reported p-value was calculated; Both weighted and unweighted UniFrac were calculated; weighted UniFrac is calculated to be p = 0.398 while unweighted UniFrac was P<0.03; Base mean abundance = 0.03 — Differential abundance of Staphylococcus aureus in the stoma calculated by Log2 fold change (y-axis) versus base mean abundance (x-axis)
Statistical Analysis 2: Comparison: Stoma Microbiota vs Healthy Thigh Skin Microbiota; Test type: Other — In this study, dissimilarities between the stomal and healthy thigh skins were tested. Observational study. Used only for visualizing trends in the data; p < 0.005, Bray-Curtis dissimilarities — Each stomal community type was distinguished by both its diversity and taxonomic composition; Nonmetric multidimensional scaling (NMDS) of Bray-Curtis dissimilarities; PERMANOVA = 0.001; Loess Regression was used to visualize temporal trends in the Shannnon Diversity and relative abundance of microbes (Staphylococcus, Streptococcus, Corynebacterium, and obligate anaerobes)

2. Secondary Outcome: Time to Equilibrium of the Bacterial Community Types Over the Duration of the Study
Description: Times required to reach stable Bacterial Community Types (CT) after the Stage 2 surgery. Dirichlet multinomial mixture modeling was used to examine the heterogeneity and optimal number of the community compositions within each sample site. Often, skin samples clustered optimally to a single community type. Five community types (CT1-5) were identified: CT1 was defined by mixed communities of obligate anaerobes. CT2 was defined as those with median Shannon diversity index of ~4.5. CT3 was defined as the microbial community with the Shannon index of ~ 0.6 and dominated by Streptococcus. CT4 and CT5 were characterized by high relative abundances of Corynebacterium (median = 49%) and Staphylococcus (median = 34%), respectively. Patients, post-surgery, stabilized to one of CT1 - CT5 stomal microbiota.
Time Frame: as for outcome 1
Population: Ten unilateral transfemoral amputees with a percutaneous osseointegrated prosthetic docking system.
Measure: Mean (Standard Deviation); unit: Months
Groups:
- Time to Reach a Stable Stomal Community Type: Overall, five Bacterial Community Types (CT1-5) were found to be present in the stomata at selected time points. These microbiota were generally temporarily unstable but with increasing time, following the Stage 2 surgery, some patients trended to a single Bacterial Community Type which was consistent until the end of the study (equilibrium).
Arm/Group | Time to Reach a Stable Stomal Community Type
Number analyzed (Participants) | 10
Months | 2.7 (2.5)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- POP 10 Patient Cohort: Patients implanted with POP devices
Arm/Group | POP 10 Patient Cohort
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
This is an observational study limited by the small number of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT02564432/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT02564432/Prot_SAP_001.pdf